CLINICAL TRIAL: NCT05714254
Title: A Randomised, Double-blind, Placebo-controlled Study of the Safety, Tolerability, and Pharmacokinetics of Multiple Ascending Doses of MEDI0618 in Healthy Male and Female Volunteers
Brief Title: Multiple Dose Study of Safety and Pharmacokinetics of MEDI0618 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: D7060C00002
Record Dates: First submitted 2022-12-12; First posted 2023-02-06 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Protocol designed to evaluate safety, tolerability and pharmacokinetic profile of an intervention for treating chronic pain
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEDI0618 (Active Comparator): A human immunoglobulin antibody to the Protease Activated Receptor 2 (PAR2)
  Interventions: Drug: MEDI0618
- Placebo (Placebo Comparator): Histidine/histidine HCl, sucrose and polysorbate
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MEDI0618 — Four doses of 100 mg IV, 200 mg IV or 200 mg SC MEDI0618 administered once every two weeks.
  Other Names: Protease-Activated Receptor 2 Antagonist
  Arms: MEDI0618
Drug: Placebo — Four doses of IV placebo or SC placebo administered once every two weeks.
  Arms: Placebo

SUMMARY:
This is a single centre, randomised, double-blind, placebo-controlled, multiple ascending dose study of MEDI0618 in healthy male and female volunteers.

Subjects will receive MEDI0618 or placebo administered by intravenous infusion or subcutaneous injection.

Safety, tolerability and pharmacokinetics of multiple ascending doses of MEDI0618 will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women of non-child bearing potential
* Aged 18 to 50 years, inclusive
* Weigh more than 50 kg
* Body Mass Index between 18 to 30 kg/m2
* Healthy, in the opinion of the Principal Investigator
* Able to understand and comply with the protocol requirements

Exclusion Criteria:

* Participation in another clinical study with a study drug within 5 half-lives of that study drug or within 3 months prior to screening, whichever is longer
* Donation of blood or plasma within 2 months prior to screening and until after the final follow-up visit
* Poor venous access
* History of severe allergy/hypersensitivity reactions or history of hypersensitivity to immunisations, immunoglobulins or biologics
* Prescence of any clinically significant illness, such as cardiovascular, neurological, pulmonary, hepatic, renal, metabolic, gastro-intestinal, urologic, immunologic or endocrine disease or disorder
* History of cancer within 5 years of screening
* History of drug abuse
* Use of prescriptions or non-prescription medicines within 7 days or 5 half-lives, whichever is longer, prior to administration of study treatments
* Any clinical abnormality on complete physical examination, vitals signs, ECG or clinical laboratory test results at screening or between screening and randomisation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | From Screening, Day 1 to Day 113
  To characterise the safety and tolerability of MEDI0618 administered IV or SC
Incidence of abnormal vital signs | From Screening, Day 1 to Day 113
  To characterise the safety and tolerability of MEDI0618 administered IV or SC
Incidence of abnormal laboratory parameters | Day -1, Day 15, Day 29, Day 43, Day 57, Day 71, Day 99, Day 113
  To characterise the safety and tolerability of MEDI0618 administered IV or SC

SECONDARY OUTCOMES:
Time to maximum observed plasma concentration (Tmax) of MEDI0618 | Day 1 to Day 113
  To characterise the pharmacokinetic (PK) profile of MEDI0618 administered IV or SC
Maximum observed plasma concentration (Cmax) of MEDI0618 | Day 1 to Day 113
  To characterise the pharmacokinetic (PK) profile of MEDI0618 administered IV or SC
Area under plasma concentration-time curve over dosing interval (AUC[tau]) of MEDI0618 | Day 1 to Day 113
  To characterise the pharmacokinetic (PK) profile of MEDI0618 administered IV or SC
Pre-dose trough concentration (Ctrough) of MEDI0618 | Day 1 to Day 113
  To characterise the pharmacokinetic (PK) profile of MEDI0618 administered IV or SC
The volume of plasma cleared of drug per unit time (CL) of MEDI0618 | Day 1 to Day 113
  To characterise the pharmacokinetic (PK) profile of MEDI0618 administered IV or SC
Anti-drug antibodies (ADA) | Day 1, Day 8, Day 29, Day 43, Day 57, Day 71, Day 99, Day 113
  To characterise the immunogenicity of MEDI0618 administered IV or SC

CONTACTS AND LOCATIONS:
Overall Officials: Stanislav Ignatenko, Principal Investigator — Charite Research Organisation, Berlin Germany
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No